CLINICAL TRIAL: NCT05007886
Title: Remote Evaluation of the Naída CI M90 (Marvel) Sound Processor
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sophie McKenny, Clinical Researcher, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 292396
Record Dates: First submitted 2021-07-28; First posted 2021-08-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Cochlear Hearing Loss; Hearing Loss
Keywords: cochlear implant; Advanced Bionics Marvel Processor
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Within-subject comparison. Remotely Evaluating latest Advanced Bionics Marvel Sound Processor for cochlear implants, from two adult groups.

DETAILED DESCRIPTION:
Within-subject comparison, standard of care CE marked Advanced Bionics device. Remote Evaluation of new CI Naida M sound processor through speech understanding in quiet and noise using standard clinical tests, subjective feedback on sound quality for a set of listening situations reflecting everyday use and a ease of use questionnaire. Two adult groups, one CI users and the other bimodal users. All tests completed remotely.

ELIGIBILITY:
Inclusion Criteria:

* CI users with a CI, HiRes90K (Advantage) or HiRes Ultra cochlear implant system
* Unilaterally implanted recipients using only a Naída Q sound processor
* Bimodal users: additionally using hearing aid on their contralateral ear

  * Minimum of 18 years of age
  * Minimum of five years' experience with their Naída Q sound processor
  * Minimum of six months experience with their contralateral hearing aid (if applicable)
  * Ability to give feedback on sound quality
  * Speech intelligibility with the BKB sentence test in noise at a +10 dB SNR > 10% as obtained during previous visits in the clinical routine or BKB >50% in quiet conditions if noise has previously not been tested
  * Fluent in English language

Exclusion Criteria:

* Difficulties additional to hearing impairment that would interfere with the study procedures
* Concurrent participation in any other clinical hearing study
* Not due to have their sound processor upgraded in line with normal clinical procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Advanced Bionics cochlear implant users due for a sound processor upgrade in line with normal standard of care. Able to access the internet and undertake tests remotely.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate difference in speech perception in noise with Naida M (Marvel) and Naida Q hearing devices | 12 months
  Understanding speech in presence of completing noise and quiet testing remotely through use of Gorilla software. This will be done through a percentage score calculated within the Gorilla software.

SECONDARY OUTCOMES:
Differences in sound clarity and comfort with Naida M (Marvel) device when listening to speech | 12 months
  Assessment in quiet, background, speech babble, household noises, traffic noise, cafeteria noise and louder alarm signals.This will be done through a measurement of specific questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge Biomedical Campus, Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No